CLINICAL TRIAL: NCT01446835
Title: Asian Clinical Evaluation of an Investigational Contact Lens for Cosmetic Effect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: P-418-C-003
Record Dates: First submitted 2011-10-03; First posted 2011-10-05 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-01

CONDITIONS: Cosmetic Appearance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- nelfilcon A (Experimental): Nelfilcon A printed contact lens randomly assigned to one eye, with etafilcon A printed contact lens assigned to the fellow eye for contralateral wear. Lenses will be worn for 20 minutes.
  Interventions: Device: nelfilcon A contact lens with print
- etafilcon A (Active Comparator): Etafilcon A printed contact lens randomly assigned to one eye, with nelfilcon A printed contact lens assigned to the fellow eye for contralateral wear.
  Interventions: Device: etafilcon A contact lens with print

INTERVENTIONS:
Device: nelfilcon A contact lens with print — Investigational spherical contact lens
  Arms: nelfilcon A
Device: etafilcon A contact lens with print — Commercially marketed (Singapore) spherical contact lens
  Other Names: 1-DAY ACUVUE DEFINE Vivid Style
  Arms: etafilcon A

SUMMARY:
The purpose of this study is to compare the cosmetic appearance of two different contact lenses on Asian eyes.

DETAILED DESCRIPTION:
Participants will be asked to evaluate the cosmetic appearance of two different contact lenses worn contralaterally for 20 minutes. No vision or comfort variables will be assessed in this cosmetic appearance and lens fit non-dispensing study.

ELIGIBILITY:
Inclusion Criteria:

* Female between 18 and 30 years of age (inclusive).
* If under 21 years of age, subject must sign informed assent and have written consent of parent or guardian to participate.
* Sign written Informed Consent.
* Chinese, Japanese, or Korean descent.
* Brown eye color.
* Spherical equivalent refractive error of -0.50 diopter (D) and between (-1.50 to -2.50D), (-3.50 to -4.50D) and (-5.50 to -6.50D).
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Eye injury or surgery within twelve weeks prior to enrollment.
* Pre-existing ocular irritation that would preclude contact lens fitting.
* Currently enrolled in any clinical ophthalmic trial.
* Evidence of systemic or ocular abnormality, infection or disease which is likely to affect successful wear of contact lenses or use of accessory solutions as determined by the investigator.
* Any use of medications for which contact lens wear could be contraindicated as determined by the investigator.
* Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 151 (Actual)
Dates: Start 2011-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Cosmetic Appearance Preference | After 20 minutes of wear
  Participant will be asked on a questionnaire, "Which lens do you prefer for looking more natural?" Subject will record on the questionnaire, "Left lens," "Right lens," or "No preference."

SECONDARY OUTCOMES:
Lens Centration | After insertion and before 20 minutes of wear
  Investigator will assess lens centration using a biomicroscope, which magnifies the appearance of the contact lens on the participant's eye. Lens centration will be graded on a 5-point scale, with 0 being centered and 4 being severe decentration with corneal exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Danny Sim Chek Hoo, B Optom (Hons), Principal Investigator — Singapore Polytechnic
Locations (1):
- Singapore Polytechnic, Spoc, W115, Singapore